CLINICAL TRIAL: NCT07346300
Title: Pediatric Physical Activity: Tailored Intervention for Children Born to Mothers With Obesity
Brief Title: We-Move With Windy: Gross Motor Development for Early Childhood
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Taren Swindle, Associate Professor, Arkansas Children's Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 260646
Record Dates: First submitted 2025-12-04; First posted 2026-01-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Physical Activities
Keywords: Preschool children; Early childhood; Physical activity intervention; Gross motor skills; Motor development
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- We Move with Windy (Experimental): Children and their moms attend 18 weeks of intervention. The first 6 weeks are fully in person for 1 hour, twice per week. The next 6 weeks are 1 in person 1 hour session and 1 zoom-based session for. The final 6 weeks are 2 sessions per week via zoom for 30-45 minuets with one in person session every other week to maintain engagement. The third phase includes home-based activity suggestions.
  Interventions: Behavioral: We Move with Windy
- Control (No Intervention): Children are encouraged to follow the physical activity recommendations of their physician.

INTERVENTIONS:
Behavioral: We Move with Windy — The intervention is an 18-week, family-centered program designed to increase physical activity and gross motor skills in preschool children born to mothers with obesity. Families in the treatment group participate in fun, developmentally appropriate movement activities-such as jumping, balancing, and throwing-through a mix of in-person sessions and technology-delivered activities that can be done at home. Activities are tailored to each child's skill level and each family's environment. Parents learn simple ways to support activity and practice skills in daily routines. Each in-person session also includes a brief fruit-and-vegetable exposure activity and recipe to promote healthy eating habits
  Arms: We Move with Windy

SUMMARY:
The long-term goal of this project is to learn whether a tailored physical activity program is practical, enjoyable, and helpful for families, and whether it has the potential to improve children's physical development and health. Before launching a large study, the research team completed several early phases to make sure the program met families' needs. First, a needs assessment was conducted with mothers to understand barriers to physical activity and what types of support would be most useful. Using this feedback, the program was refined and tested with three mother-child pairs over six weeks. Finally, there was an 18-week pilot randomized trial to examine feasibility and acceptability.

Researchers are now conducting a larger randomized trial with up to 266 families. Half of the families are randomly assigned to receive the physical activity program, and half to a comparison group. The program combines fun, age-appropriate movement activities for children with practical support for parents. Sessions focus on building core movement skills such as jumping, balancing, running, and throwing, while also encouraging confidence, coordination, and enjoyment of being active. Activities can be adapted to each child's ability and home environment, making the program realistic for busy families.

The program includes both in-person sessions and technology-based activities. In-person sessions provide hands-on support for learning new skills. Technology-based activities offer simple ideas families can use at home or during daily routines, such as hopping games, balance challenges, or quick movement breaks.

Because parents in earlier phases wanted nutrition support, in-person sessions also includes a brief, child-friendly exposure to fruits and vegetables, along with simple recipes. A "Tasting Party" at the start of the program allows children to try different foods, and Veggie Meter scans at the beginning and end of the study help track changes in fruit and vegetable intake.

Overall, this study will help determine whether a family-tailored physical activity program is a promising approach to improving physical activity, movement skills, and early health indicators in young children born to mothers with obesity.

DETAILED DESCRIPTION:
Children born to mothers with obesity are at elevated risk for obesity and related cardiometabolic conditions beginning early in life. Evidence suggests that these children may engage in lower levels of physical activity, experience delays in gross motor skill development, and encounter additional barriers to movement and active play prior to school entry. Early childhood represents a critical window for establishing movement competence, physical activity behaviors, and dietary exposures that track into later childhood and adulthood. Interventions during this developmental period may therefore offer an important opportunity to reduce health risk trajectories. To address this need, the research team developed a family-based, developmentally tailored physical activity intervention designed to support gross motor skill development, promote enjoyable movement experiences, and reinforce healthy eating behaviors among preschool-aged children at elevated risk.

Prior to initiating the this trial, the team conducted a series of formative and pilot phases to refine intervention components and ensure alignment with family needs and preferences. First, a needs assessment with mothers of preschool-aged children was conducted to identify perceived barriers to child physical activity, contextual constraints within the home environment, and desired forms of support. Findings from this phase informed iterative refinement of program content and delivery strategies. Next, the revised materials were pre-tested with three mother-child dyads over a six-week period to assess usability, engagement, and logistical feasibility. Building on these findings, we conducted an 18-week pilot randomized trial to further evaluate feasibility, acceptability, and preliminary implementation outcomes.

The current study is a larger-scale randomized controlled trial enrolling up to 266 families. Families are randomized to either the intervention condition or a control condition. The intervention integrates developmentally appropriate, play-based movement activities for children with structured support for parents to facilitate and reinforce physical activity in the home. Intervention sessions focus on foundational gross motor skills-including jumping, balancing, running, and throwing-while also fostering coordination, self-efficacy, and positive affect toward physical activity. Activities are designed to be adaptable to children's developmental skill levels and household environments, enhancing feasibility for diverse families.

Intervention delivery combines in-person and technology-delivered components. In-person sessions provide hands-on instruction and guided practice to support skill acquisition and movement confidence. Technology-delivered components extend learning beyond in-person sessions by offering brief, low-burden activity prompts that families can integrate into daily routines (e.g., movement games during transitions, short balance or hopping challenges, or active play during household tasks). This hybrid approach is intended to promote skill generalization, reinforce parent engagement, and support sustained physical activity opportunities in the home.

In response to strong interest expressed by parents during formative work, nutrition exposure is embedded in in-person sessions. Children participate in brief, developmentally appropriate fruit and vegetable tastings, accompanied by simple, family-friendly recipes to encourage at-home practice. Objective assessment of fruit and vegetable intake is conducted at baseline and follow-up using Veggie Meter scans to examine changes in carotenoid status over time.

Across all phases, the intervention is grounded in the principle that young children learn most effectively through positive experiences, encouragement, repetition, and opportunities for mastery. Because caregivers-particularly mothers-play a central role in shaping home routines and modeling health behaviors, the intervention targets the family unit rather than the child alone. Primary outcomes for the trial include feasibility, acceptability, and fidelity of intervention delivery, as well as child-level changes in physical activity, gross motor skill development, and early health indicators. Findings from this study will inform the potential of a family-tailored physical activity intervention to alter early-life health trajectories among children born to mothers with obesity.

*The study was registered once the requirement for registration in an ICMJE-accepted registry was identified. No changes were made to study procedures or participant activities as a result of this timing.

ELIGIBILITY:
Inclusion Criteria: Mother-child pair where the mother has

* Body mass index >30 and
* The child is between 3 and 5 years of age.

Exclusion Criteria:

* mothers sharing that a doctor has requested that either mother or child not exercise (e.g., asthma).

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Test of Gross Motor Development-2 | At baseline (prior to intervention initiation) and at post-intervention (approximately 19-25 weeks after baseline).
  The Test of Gross Motor Development-2 (TGMD-2)31 was used to assess children's motor skill competence. The TGMD-2 assesses 12 skills: run, gallop, hop, leap, horizontal jump, slide (locomotor skills); striking a stationary ball, stationary dribble, kick, catch, overhand throw, and underhand roll (object control skills). A research team member demonstrates the proficient technique to the child; then, the child is asked to perform the skill twice. Researchers score each attempt to perform the skill based on set criteria. Scores on the TGMD range from 0 to 100 with higher scores reflecting greater gross motor skill proficiency.

SECONDARY OUTCOMES:
Raman Spectroscopy | At baseline (prior to intervention initiation) and at post-intervention (approximately 19-25 weeks after baseline).
  The Veggie Meter uses Raman Spectroscopy (RS) technology to measures skin carotenoid levels as a biomarker for colorful FV intake with an optical hand scan. RS reflects intake over the prior 4 weeks and is sensitive to individual differences and experimental changes. Children are asked to use hand sanitizer prior to placing their finger in the RS scanner. Scores range from 0 to 100 with higher scores reflecting greater carotenoid intake.
Accelerometry | One 7-day assessment period during the intervention (approximately weeks 6-12) and one 7-day assessment period at post-intervention (approximately 19-25 weeks)
  Staff provide accelerometer equipment and instructions to family and gather the equipment at the next scheduled on-site intervention assessment. Participants wear the monitors for up to 8 days, including two weekend days, only removing them during showers/baths and water activities such as swimming in a pool, lake, going to a water park, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Taren Swindle, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Research Institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No